CLINICAL TRIAL: NCT07125768
Title: Comparative Study Between Thermal Radiofrequency Neurolysis Versus Alcoholic Neurolysis of the Genicular Nerves for Treatment of Chronic Knee Pain in Advanced Knee Osteoarthritis
Brief Title: Thermal Radiofrequency Neurolysis Versus Alcoholic Neurolysis of the Genicular Nerves for Treatment of Chronic Knee Pain in Advanced Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hesham Mahmoud Elsayed Eldamhogy, Resident of Anesthesiology, Surgical Intensive Care and Pain Management Department, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS603/5/24
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Thermal Radiofrequency Neurolysis; Alcoholic Neurolysis; Genicular Nerves; Treatment; Chronic Knee Pain; Advanced Knee Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients received C-arm guided neurolysis of superior medial [SM], superior lateral [SL], and inferior medial [IM] genicular nerves by thermal radiofrequency.
  Interventions: Other: Thermal Radiofrequency Neurolysis
- Group II (Active Comparator): Patients received C-arm guided injection of each of the three genicular nerves with 1 ml of a solution containing 70% alcohol in 0.25% lidocaine.
  Interventions: Other: Alcoholic Neurolysis

INTERVENTIONS:
Other: Thermal Radiofrequency Neurolysis — Patients received C-arm guided neurolysis of superior medial [SM], superior lateral [SL], and inferior medial [IM] genicular nerves by thermal radiofrequency.
  Arms: Group I
Other: Alcoholic Neurolysis — Patients received C-arm guided injection of each of the three genicular nerves with 1 ml of a solution containing 70% alcohol in 0.25% lidocaine.
  Arms: Group II

SUMMARY:
This study aimed to compare the strength and duration of pain relief, quality of life and analgesic consumption between patients who undergo conventional thermal radiofrequency vs patients who undergo chemical neurolysis on genicular nerves by alcohol in chronic knee osteoarthritis pain.

DETAILED DESCRIPTION:
Knee osteoarthritis is a degenerative joint disease characterized by the degradation of the articular cartilage, with many factors implicated in the disease pathogenesis.

Chronic pain of knee osteoarthritis is a common clinical symptom leading to restricted movement, disability, psychological distress, and impaired quality of life.

The targeted genicular nerves are those that had a close topographic relationship with the bone cortical surfaces, such as the femoral epicondyles (Superior medial [SM] and Superior lateral [SL] genicular nerves) and the medial tibial epicondyle (Inferior medial [IM] genicular nerve).

Nerve ablation causes iatrogenic neural degeneration, aiming only for sensory or sympathetic denervation without motor deficits. The nerve ablation methods currently available are performed by either thermal ablation using radiofrequency or chemical ablation using alcohol or phenol.

Chemical neurolysis techniques can be an effective method to accomplish a larger, more thorough lesioning than radiofrequency ablation and are capable of covering the anatomical variability of genicular nerves, so ensuring a better success rate and outcome with less cost and less logistic support.

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 60 years.
* Both sexes.
* Stage 3 and 4 knee osteoarthritis in patients who aren't responding to pharmacological treatment and aren't good candidates for knee replacement surgery.

Exclusion Criteria:

* Neurological disorders (Previous cerebrovascular stroke, neuropathy, or weakness).
* Bleeding disorders.
* Infection at or near the injection site.
* Presence of a pacemaker or defibrillator.
* Acute knee injury.
* Unstable knee joint.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Improvement of knee osteoarthritis pain | 6 months post-procedure
  Improvement of knee osteoarthritis pain according to Visual Analogue Scale (VAS). VAS: which was a subjective scale used to quantitatively assess pain (0 = No pain, 10 = Severe pain).

SECONDARY OUTCOMES:
Improvement of quality of life | 6 months post-procedure
  Improvement of quality of life according to Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score. WOMAC is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscale areas: Each scale uses the following descriptors for all items: none, mild moderate, severe, and extreme. These correspond to an ordinal scale of 0-4. The scores were summed up for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68.
Decrease of analgesic requirements of pain control after neurolysis. | 6 months post-procedure
  All patients received standard analgesic regimen in the form of non-steroidal anti-inflammatory drugs (Diclofenac Sodium) until they reach the same satisfactory level of pain control, and we asked the patient to use diary to record the amount of analgesia used during the follow up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of the study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of the study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.